CLINICAL TRIAL: NCT04132687
Title: To Determine the Efficacy of Autologous Blood Patch Therapy in Reducing Air Leak in Secondary Spontaneous Pneumothorax: A Proof-of-Concept Study
Brief Title: ABPT in Secondary Pneumothorax With Persistent Airleak Study
Acronym: ABPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ngai Chun Li, Principal Investigator, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABPT_protocol_version 3_0
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Autologous Blood Patch Therapy
Keywords: digital chest drain device

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- autologous blood patch (Other): autologoust blood patch therapy
  Interventions: Procedure: autologous blood patch therapy

INTERVENTIONS:
Procedure: autologous blood patch therapy — use autologous blood as blood patch therapy in persistent air leak

SUMMARY:
This is a prospective clinical trial with each patient serving as his/her own control. Patients will be recruited in three different Hong Kong hospital. All patients at the recruitment centers with ongoing air leak after ≥ 3 days from the initial diagnosis of SSP will be approached by site investigators. Patient consented to enter the study will have their rate of air leak measured on day 3 (or after if enrolled later than day 3) byreplacing the conventional chest drain system with the digital chest drainage device (Thopaz).

Autologous blood patch will be instilled if the patient still has persistent air leak on day 5 of chest drain insertion ( or 48 hours of electronic chest drain measurement of airleak).

DETAILED DESCRIPTION:
The patient must have a chest tube in place and checked to be patent. Approximately 1.5ml/kg of venous blood will be withdrawn from the patient and immediately instilled it into the pleural cavity with aseptic technique via the chest tube already in situ. (There is no standard amount of blood used for ABPT. A small randomized study advocated that the use of 1.5ml/kg as it provided the optimal benefits.) The drain is then flushed with 20ml normal saline to avoid clotting. The tube of the drain is immediately elevated to 60cm above the insertion point of the chest tube at the patient's chest wall for 2 hours. This method allows ongoing evacuation of any air leak while the instilled blood can stay within the pleural cavity. The tube is never clamped at any stage to avoid any risk of tension pneumothorax. The patient was asked to change his position in bed every 10 minutes (supine, right lateral, prone, left lateral, head down and sit upright) during the two-hour period to aid distribution of blood over the visceral pleura. The tube is returned to normal position after two hours and the patient is free to ambulate. Analgesia is freely available for the patient should the need arise, but will not be prescribed routinely as existing data suggest it is uncommon.

Patients will remain under close observation after the instillation for the next 6 hours by experienced respiratory doctors and nurses, in particular for any suggestion of tube blockage or worsening pneumothorax. The tube will be flushed with saline (of an amount similar to the dead space of the tube) if that occurs. In the very unlikely event that the blockage is not correctable, a new chest tube may be placed if deemed clinically necessary. Prophylactic antibiotics will be given at the discretion of the attending clinician. The amount of air leak is measured continuously before and after ABPT using Thopaz system. Patients are free to receive any other therapy (except pleurodesis) during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older;
* radiographically proven pneumothorax and underlying lung disease (either pre-existing or shown in diagnostic imaging at presentation);
* chest tube inserted which still shows an air leak at day 5 (or later) after the first radiographic evidence of a pneumothorax.

Exclusion Criteria:

* inability to provide informed consent;
* a chest tube smaller than 12 F (because of the risk of blockage by blood)
* bilateral pneumothorax
* uncorrectable coagulopathy
* active or recent (within 6 weeks) pleural infection
* use of long term steroid or immunosuppressant
* septicaemia or active extrapleural infection (eg pneumonia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
air leak reduction | 48 hours
  percentage of air leak reduction after autologous blood patch

CONTACTS AND LOCATIONS:
Overall Officials: Chun Li Dr Ngai, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No